CLINICAL TRIAL: NCT06826820
Title: Fertility: Infection and Inflammation
Acronym: InFert
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 34-459
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Observational Study of IVF Patients
Keywords: IVF; follicular fluid; blood samples

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, follicular fluid, cells (blood cells, granulosa cells), media for embryo culture, ejaculate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing IVF treatment: no intervention

SUMMARY:
The investigators explore whether inflammatory factors and infections in collected samples are altered in fertility issues and if they can predict pregnancy outcomes. The investigators focus on pro- and anti-inflammatory markers, such as cytokines, metabolic parameters (e.g., blood lipids, hormones, bile acids), and viral infections (e.g., HPV, herpesviruses). A standard blood panel is also performed.

Fertility issues are rising due to aging, infections, environmental toxins, and lifestyle factors (e.g., BMI, diabetes). Fertilization and implantation involve complex interactions between the egg, sperm, embryo, and endometrium, which can be disrupted by inflammatory processes from infections, metabolic imbalances, or environmental toxins. IVF allows access to unique samples that help identify these processes and their impact on fertility.

1. Sample Collection & Analysis

   * Diagnostic Cycle: Blood samples (early/late follicular phase), endometrial sample (7 days post-ovulation), and body composition analysis (BOD POD).
   * Oocyte Retrieval: Blood, follicular fluid, vaginal swab, and another body composition analysis (BOD POD). The male partner provides blood and an ejaculate sample.
   * After IVF: The culture medium where the fertilized egg grows is collected. Samples are analyzed for hormones, cytokines, metabolites, nucleic acids, proteins, and immune cells. Some granulosa cells are isolated and cultured.
2. Clinical & Fertility Parameters

   The main outcome is a clinical pregnancy, but additional factors are examined:
   * Patient: IVF reason, AMH levels, pre-existing conditions, medications, smoking, pregnancy duration.
   * IVF parameters: Follicle counts, retrieved oocytes, fertilization method (IVF/ICSI), embryo quality, implantation rate, miscarriage rate, and live birth rate.
   * Newborn: Birth weight, length, sex.
3. Control Groups & Data Management Control groups consist of couples where infertility is attributed to only one partner. All samples are pseudonymized before analysis to ensure data privacy.

DETAILED DESCRIPTION:
The investigators aim to investigate whether inflammatory and inflammation-inducing factors detectable in the collected samples, as well as infections present in these samples, are altered in cases of fertility issues and whether these factors could be predictive of pregnancy progression and child outcomes. Specifically, factors that mediate inflammation-acting either pro-inflammatory or anti-inflammatory-will be examined for their association with pregnancy establishment. This includes, for example, signaling molecules such as cytokines, metabolic and endocrinological parameters that may contribute to a pro-inflammatory milieu (e.g., hyperglycemia, blood lipids, hormones), viral infections that may influence fertility (e.g., human papillomavirus (HPV), herpesviruses). Additionally, a standard blood panel will be performed.

Fertility issues are increasing in both women and men. The causes are not only due to the higher age of couples wishing to conceive but also to infections, environmental factors (e.g., environmental toxins), and lifestyle-associated factors (e.g., BMI, increased body fat percentage, and diabetes). The fertilization of the egg and the implantation of the embryo into the endometrium is a highly complex process influenced by many factors. The egg, sperm, embryo, and endometrium all play a crucial role. Essential are, on the one hand, factors secreted by these components, which are present in maternal blood, follicular fluid, or ejaculate, and on the other hand, factors produced by the mother that influence the egg, fertilization, embryo, and endometrium.

Inflammatory processes, such as those occurring due to viral or bacterial infections, metabolic dysregulations (diabetes or obesity), or exposure to environmental substances (environmental toxins), may alter the normal milieu and thereby affect fertilization and implantation. In the context of assisted reproductive technologies (in vitro fertilization, IVF), the investigators have the opportunity to analyze samples that are not accessible during natural conception. These samples allow us to identify the presence of inflammatory processes and investigate their impact on pregnancy establishment.

1. Sample Collection:

   In the diagnostic cycle-a cycle preceding further fertility treatment, during which possible causes of infertility are assessed-blood samples in both the early and late follicular phase (cycle days 2-5 and 19-21) will be collected and an endometrial sample (7 days after ovulation). Additionally body composition (including body fat percentage) is measured in the BOD POD and via ultrasound.

   During oocyte retrieval, the investigators collect blood, follicular fluid (individually the primordial follicle, the rest pooled, and a microbiological vaginal swab. Moreover, body composition is again measured in the BOD POD. From the male partner the investigators collect a blood sample and an aliquot of the ejaculate.

   After in vitro fertilization (IVF), the culture medium in which the fertilized egg develops into a blastocyst is collected.
2. Sample Analysis:

In blood samples and follicular fluid, the investigators will analyze signaling molecules (hormones, cytokines, etc.), Metabolites (including amino acids, bile acids), Proteins, RNA molecules, cell-free DNA, oligosaccharides, and immune cells. For some follicular fluid samples, granulosa cells will be separated by centrifugation and cultured. Body composition/% body fat will be measured.

The main readout is the establishment of a clinical pregnancy. However, additional clinical information about the patient is also considered, including reason for IVF treatment, diagnosis, relevant pre-existing conditions, surgeries, or long-term medication use, smoking status, anti-Müllerian hormone (AMH) levels, stimulation protocol, duration of pregnancy. Furthermore, clinical information about the neonate is collected, including birth weight, birth length, and sex.

Additionally, the following fertility diagnostic parameters are documented and analyzed: Antral follicle count (AFC), number of preovulatory follicles, number of follicles on the day of oocyte retrieval, number of retrieved oocytes, follicular Output Rate (FORT), follicle-to-Oocyte Index (FOI), oocyte utilization rate, oocyte maturation status (MII, MI, GV, zona pellucida), fertilization method (IVF, ICSI), pronucleus classification (PN1-4), fertilization rate, mnumber of blastocysts, blastocyst morphology, blastocyst formation rate, eEmbryo quality, fresh or frozen embryo transfer, implantation rate, biochemical pregnancy rate, miscarriage rate, live birth rate.

Experimental parameters will be evaluated using clinical findings to gain a comprehensive understanding of patient fertility, response to IVF treatment, and, if applicable, pregnancy progression.

Control Groups The control group consists of samples from couples in whom infertility is attributed solely to the male partner (serving as a control for female patient samples) or solely to the female partner (serving as a control for male partner samples).

All samples are pseudonymized by research nurses before analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women, and optionally their partners, aged 18 or older with written consent to participate in the study.

Exclusion Criteria:

* Minors and patients unable to provide consent. Conditions or circumstances that, in the opinion of the investigator or treating physician, could interfere with the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women (and optionally partners) undergoing IVF treamtent
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2032-12-20 (Estimated); Study Completion 2032-12-20 (Estimated)

PRIMARY OUTCOMES:
clincal pregnancy | 7 weeks after oocyte transfer
  establishment of a clinical pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided